CLINICAL TRIAL: NCT05144828
Title: Efficacy of Intercostal CryoAnalgesia in Patients Undergoing Robot Assisted Anatomic Lung Resection
Brief Title: Efficacy of Intercostal CryoAnalgesia in Robotic Lung Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Mario Gasparri, MD, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO40665
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Pain, Postoperative; Lung Diseases
Keywords: Atricure; CryoNB; cryoanalgesia; Medical College of Wisconsin
MeSH Terms: conditions — Pain, Postoperative; Lung Diseases | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intercostal Nerve Cryoablation plus Standard of Care (SOC) Pain Control (Experimental): Intercostal nerve cryoablation using the CryoICE® CRYOS-L cryoablation probe and an intercostal nerve block of nerves 4-9 performed using 0.5% Marcaine with Epinephrine plus prescribed post-operative pain medication, including tramadol, tylenol, and robaxin
  Interventions: Device: Intercostal Nerve Cryoablation; Drug: Patient-controlled analgesia (PCA)
- Standard of Care (SOC) Pain Control (Active Comparator): Intercostal nerve block of nerves 4-9 using 0.5% Marcaine with Epinephrine plus prescribed post-operative pain medication, including tramadol, tylenol, and robaxin
  Interventions: Drug: Patient-controlled analgesia (PCA)

INTERVENTIONS:
Device: Intercostal Nerve Cryoablation — Patients will receive intraoperative intercostal nerve cryoablation using CryoICE® CRYOS-L cryoablation probes (AtriCure, Inc) to intercostal spaces 4th to 10th in thoracoabdominal aortic repairs and 4th to 8th in descending thoracic aortic repair cases prior to wound closure.
  Other Names: CryoICE CRYOS-L cryoablation probes (Atricure, Inc.)
  Arms: Intercostal Nerve Cryoablation plus Standard of Care (SOC) Pain Control
Drug: Patient-controlled analgesia (PCA) — Patients will have access to the standard PCA (patient-controlled analgesia) offered at Froedtert Hospital. This includes tylenol 650 mg oral, robaxin 500 mg oral, and tramadol 25-50 mg oral. All patients will have the first two ports placed at which time an intercostal nerve block of nerves 4-9 will be performed using 0.5% Marcaine with Epinephrine.

SUMMARY:
This is a single center, single surgeon, prospective, randomized trial examining the addition of Cryo Nerve Block during robot assisted thoracoscopic anatomic lung resection surgery

DETAILED DESCRIPTION:
Thoracic surgical procedures are consistently reported to be among the most painful surgical incisions currently used. Trauma to the skin, muscle, intercostal nerves, bones and pleura all contribute and lead to activation of various pain pathways including somatic, visceral, neurogenic and phrenic. In the short term, this pain leads to ineffective cough and pulmonary hygiene resulting in respiratory complications and prolonged hospital stays while in the longer term it leads to prolonged recovery, delayed return to work and in some instances, chronic post thoracotomy pain syndromes. Minimally invasive approaches such as standard thoracoscopy or robotic assisted thoracoscopy have certainly decreased some of this trauma as evidenced by decreased length of stays and decreased complication rates however even with these minimally invasive techniques, recovery to 80% of baseline is 25 days and 9.4% of patients are still using narcotics after 90-180 days.

Several options are available in the management of pain following thoracic surgery with a multimodal pain medicine approach being most common. Opioids, unfortunately, are a relatively large part of this approach and are often relied upon despite their relatively unfavorable adverse event profile and risk for addiction. Many of the other pain adjuncts often used with thoracotomies such as epidural catheters or intraoperatively placed pain catheters are not really reasonable when using minimally invasive approaches as the hospital length of stay is 1-2 days. Intercostal cryoanalgesia has been shown to be a safe and effective strategy for postoperative pain management in patients undergoing thoracotomy. Recent studies have demonstrated the beneficial effect of cryoanalgesia for post-thoracotomy pain in reduction of opioid requirement, reduction in post-operative pain scores, and superior pulmonary function (higher FEV1 and FVC values)5 and that it can produce temporary neurolysis for up to two months without long-term histological nerve damage. To date it has not been studied when using minimally invasive techniques whether it be standard thoracoscopy or robotic assisted thoracoscopy but it would stand to reason that it would be equally or maybe more effective in this patient population and truly maximize the benefits of a minimally invasive approach.

We therefore propose to assess whether intra-operative intercostal cryoanalgesia using the cryoICE® probe provides superior post-operative analgesia as compared to our current standard pain management strategy in patients undergoing robotic assisted thoracoscopic anatomic lung resection and allows for decreased opioid use and more rapid recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* Acceptable surgical candidate
* Willing and able to return for scheduled follow-up visits

Exclusion Criteria:

* Patients undergoing or requiring conversion to thoracotomy
* Patients with chronic pain syndromes requiring treatment within the last year
* Patients with a history of illicit drug use
* Patients with a history of heavy alcohol use in the last five years as determined by the principal investigator
* Patients currently using opioids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gasparri, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control | Standard of Care (SOC) Pain Control
Started | 17 | 16
Completed | 15 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control | Standard of Care (SOC) Pain Control | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (6.3) | 65.3 (13.8) | 66.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale (VAS) Pain Score
Description: The visual analogue scale is a pain assessment tool intended to help patient care providers assess pain according to individual patient needs. A 0-10 scale is used for patient self-assessment with 0 meaning no pain and 10 meaning worst possible pain.
Time Frame: 14 Days post-operatively, day 30, day 60, day 90, day 120, day 150, day 180
Population: Daily VIS Score
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 17 | 16
scores on a scale
  Day 0 | 4.94 (2.22) | 7.50 (1.41)
  Day 1 | 4.57 (2.28) | 6.25 (1.98)
  Day 2 | 4.14 (2.51) | 5.44 (1.67)
  Day 3 | 4.36 (2.53) | 5.06 (1.88)
  Day 4 | 3.57 (2.31) | 5.00 (1.83)
  Day 5 | 3.79 (2.36) | 4.19 (2.10)
  Day 6 | 4.07 (2.50) | 3.56 (1.97)
  Day 7 | 3.57 (2.24) | 3.19 (1.76)
  Day 8 | 3.64 (2.24) | 2.94 (2.46)
  Day 9 | 2.21 (1.81) | 2.56 (2.00)
  Day 10 | 2.6 (1.50) | 2.75 (1.53)
  Day 11 | 2.67 (1.95) | 2.81 (1.64)
  Day 12 | 2.53 (1.81) | 2.50 (1.26)
  Day 13 | 2.47 (1.51) | 2.50 (1.90)
  Day 14 | 3.13 (2.20) | 2.25 (1.73)
  Day 30 | 2.29 (1.83) | 1.20 (1.57)
  Day 60 | 1.06 (1.00) | 1.27 (2.31)
  Day 90 | 0.60 (0.99) | 0.60 (1.30)
  Day 120 | 0.47 (0.92) | 0.67 (1.40)
  Day 150 | 0.33 (0.82) | 0.53 (1.55)
  Day 180 | 0.47 (0.83) | 0.67 (1.40)

2. Primary Outcome: Pain Medication Use
Description: Patients will be asked about their pain medication use daily for 21 days following surgery. Total mg of postoperative pain medication taken will be collected.
Time Frame: 21 Days post-operatively
Measure: Mean (Standard Deviation); unit: mgs
Arm/Group | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 17 | 16
mgs
  Day 0 | 6.47 (11.29) | 24.38 (16.21)
  Day 1 | 8.24 (10.89) | 23.44 (17.77)
  Day 2 | 3.00 (6.84) | 19.69 (15.65)
  Day 3 | 2.65 (6.40) | 16.25 (14.55)
  Day 4 | 2.06 (5.32) | 10.63 (13.52)
  Day 5 | 2.06 (5.32) | 9.38 (11.09)
  Day 6 | 2.94 (6.14) | 6.88 (9.29)
  Day 7 | 2.65 (4.72) | 4.69 (6.94)
  Day 8 | 3.82 (5.74) | 3.44 (6.25)
  Day 9 | 2.65 (5.34) | 3.13 (6.29)
  Day 10 | 1.76 (4.98) | 2.50 (4.83)
  Day 11 | 1.47 (3.86) | 2.50 (4.83)
  Day 12 | 1.18 (2.81) | 3.75 (6.45)
  Day 13 | 1.18 (2.19) | 3.13 (6.29)
  Day 14 | 1.18 (2.19) | 3.44 (5.98)
  Day 15 | 1.47 (3.86) | 2.19 (5.47)
  Day 16 | 1.76 (3.93) | 2.50 (5.48)
  Day 17 | 1.47 (3.86) | 1.88 (4.03)
  Day 18 | 0.88 (1.96) | 0.94 (2.72)
  Day 19 | 0.88 (1.96) | 0.94 (2.72)
  Day 20 | 1.03 (2.35) | 0.31 (1.25)
  Day 21 | 0.74 (2.12) | 0.63 (2.50)

3. Secondary Outcome: M.D. Anderson Symptom Inventory (MDASI) Score
Description: The MD Anderson Symptom Inventory (MDASI) is a multi-symptom patient-reported outcome (PRO) measure for clinical and research use. The inventory assesses severity of multiple symptoms and the impact of symptoms on daily functioning during the last 24 hours. The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 numerical rating scale, with 0 being "not present" and 10 being "as bad as you can imagine." The mean score symptom severity (of the 13 core symptom items) will be calculated with a higher score indicating a higher severity of symptoms and a lower score indicating a lower severity of symptoms.
Time Frame: Post-operative day 1, week 1, week 2, week 3, week 4, week 5, week 6
Reporting Status: Not Posted

4. Secondary Outcome: Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Score
Description: The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale is an assessment tool to analyze and classify pain. The primary purpose of this test is to assess whether the pain experienced is predominantly due to nerve damage or not. The LANSS comprises of a 7-item pain scale, including sensory descriptors and items for sensory examination. Each of the 7 items is awarded a number of points, depending on the answer choice. In general, answers like no or that signal normal function are awarded 0 points and those that signal a pain related symptom or sign are awarded a number of points varying from 1 to 5, depending on the severity of the particular sign. The final score ranges from 0 to 24. The interpretation is that patients with scores below 12 are less likely to carry a neuropathic cause for their pain whilst in the case of patients scoring 12 or more, there is a higher chance for the underlying mechanism to be neuropathic.
Time Frame: Post-operative month 1, month 3, month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: D0 (date of procedure) through D21
Arm/Group | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control | Standard of Care (SOC) Pain Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 3/17 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intercostal Nerve Cryoablation Plus Standard of Care (SOC) Pain Control (N=17) | Standard of Care (SOC) Pain Control (N=16)
Prolonged air-leak (Respiratory, thoracic and mediastinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT05144828/Prot_000.pdf